CLINICAL TRIAL: NCT00946257
Title: A Randomised, Single-blind, Placebo-controlled, Study to Evaluate the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Single Ascending Administration of Otelixizumab in Subjects With Type 1 Diabetes Mellitus
Brief Title: Subcutaneous Administration of Otelixizumab to T1DM Patients
Acronym: RAO112438
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 112438
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — otelixizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): 0.3 mg dose
  Interventions: Drug: Otelixizumab
- Cohort 2 (Experimental): 0.6 mg dose
  Interventions: Drug: Otelixizumab
- Cohort 3 (Experimental): 1.2 mg dose
  Interventions: Drug: Otelixizumab
- Cohort 4 (Experimental): 1.8 mg dose
  Interventions: Drug: Otelixizumab
- Cohort 5 (Experimental): 2.4 mg dose
  Interventions: Drug: Otelixizumab
- Cohort 6 (Experimental): 3.0 mg dose
  Interventions: Drug: Otelixizumab

INTERVENTIONS:
Drug: Otelixizumab — A humanized, aglycosyl, non-mitogenic, anti CD3 monoclonal antibody (MAb) directed against the ε domain of the human lymphocyte antigen CD3.

SUMMARY:
This study will assess the subcutaneous administration of otelixizumab to T1DM patients. The study will provide safety, tolerability, pharmacodynamic and pharmacokinetic information which will enable the identification of appropriate safe and well-tolerated subcutaneous dosage regimens to be used in subsequent clinical studies. This study will consist of a screening phase, followed by an in-house phase whereby otelixizumab will be administered to cohorts that will be staggered at each dose level.

DETAILED DESCRIPTION:
Otelixizumab is a humanized, aglycosyl, non-mitogenic, anti CD3 monoclonal antibody (MAb) directed against the ε domain of the human lymphocyte antigen CD3, which is currently undergoing phase III clinical trials in adult new-onset type I diabetes mellitus patients and has been evaluated in rheumatoid arthritis and psoriasis patients in small exploratory studies. In previous studies, otelixizumab has been administered by intravenous infusion. This study is a randomised, single-blind, placebo-controlled, study of otelixizumab administered subcutaneously in Type 1 Diabetes Mellitus (T1DM) subjects.

The assessment of otelixizumab in T1DM subjects will provide safety, tolerability, pharmacodynamic and pharmacokinetic information following subcutaneous administration which will enable the identification of appropriate safe and well-tolerated subcutaneous dosage regimens to be used in subsequent clinical studies. This study will consist of a screening phase, followed by an in-house phase whereby otelixizumab will be administered to cohorts that will be staggered at each dose level. Approximately 6 dose levels, covering up to a 10-fold dose range, will be evaluated. A single subcutaneous dose of otelixizumab will be administered on Day 1 and, serial blood samples will be obtained for clinical laboratory testing, determination of pharmacodynamic markers, serum otelixizumab PK parameters, and immunogenicity. Safety and pharmacodynamic data from the previous dose(s) will be evaluated prior to dose escalation or modification to ensure safety and to achieve target systemic peripheral blood pharmacology. Adverse events, laboratory values, vital signs and ECG's will be monitored closely during this study. All subjects in the study will undergo long-term follow-up out to 48 months to monitor and ensure patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 mIU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section TBC if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.

Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 to sufficiently minimize the risk of pregnancy. Female subjects must agree to use contraception for at least 2 weeks prior to dosing and for at least 60 days after dosing.

* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 2 weeks after dosing.
* Body weight > or = 50 kg and BMI within the range 18 - 30 kg/m2 (inclusive).
* Confirmed diagnosis of insulin-requiring T1DM according to the America Diabetes Association criteria and on a relatively stable insulin regimen, with HbAlc > or = 9%.
* Positive for at least one of the following T1DM-related autoantibodies: anti-GAD (glutamic acid decarboxylase) and/or anti IA 2A.
* Random plasma C-peptide level must be above the level of assay detection at Screen. NOTE: If the screening random plasma C-peptide level is undetectable, subjects must have a Mixed Meal Stimulated C-peptide (MMSCP) equal to or greater than 0.15 nmol/L (0.45 ng/mL) to be eligible for study participation.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Average QTcB < 450 msec.
* No history of splenectomy.
* Subject is seropositive for EBV with < 10,000 copies of EBV DNA per 106 lymphocytes as determined by quantitative polymerase chain reaction.
* CD4+ lymphocyte counts within normal limits within the 30 days before the first dose of study drug.
* Chest X-ray with negative finding at screening
* The subject has no current or prior malignancy, other than non-melanoma skin cancer (subject must have had fewer than 5 occurrences of non-melanoma skin cancer, and the last occurrence must not be within 3 months of study entry).
* Laboratory tests normal at screening or judged not clinically significant by the investigator (except for labs relating to T1DM which may include but not limited to HbA1C and glucose).

Exclusion Criteria:

* A positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines
* Positive for anti Hepatitis C antibody, Hepatitis B surface antigen, and Hepatitis B core antibody at screening
* A positive test for HIV antibody.
* A positive test for syphilis.
* History of regular alcohol consumption within 6 months of the study defined as:

an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.

* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Significant and/or active disease in any body system outside of type 1 diabetes mellitus. Examples of significant diseases include but are not limited to: coronary artery disease, congestive heart failure, uncontrolled hypertension, emphysema, seizure disorder.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* The subject has previously received otelixizumab or any other anti-CD3 Mab (e.g., OKT3, ChAglyCD3, or OKT3 ala ala) or anti-CD20 Mab (e.g. rituximab) at any time.
* Use of prescription or non-prescription drugs, except insulin, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Subjects who have had a prior allergic reaction, including anaphylaxis, to otelixizumab or any other human, humanized, chimeric, or rodent antibodies.
* History of frequent headaches and/or migraine.
* History of atopy.
* History of hypotension or orthostatic hypotension.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Subject received a vaccine within 30 days before the first dose of study drug, or requires a vaccine within 30 days after the last dose of study drug.
* Subjects who have experienced a significant systemic infection within 3 months before the first dose of study.
* Pregnant or lactating females
* The subject has clinically significant abnormal laboratory values during the screening period, other than those due to T1DM. Abnormal values are permitted if, upon re-test, the abnormality was resolved.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-07-08 (Actual); Primary Completion 2011-08-01 (Actual); Study Completion 2013-06-25 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability after a single dose of otelixizumab in T1DM patients | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Belgium (5):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Merksem

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 112438 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112438?search=study&search_terms=112438#rs
- Available data/document: Statistical Analysis Plan: 112438 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112438 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112438 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112438 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112438 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112438 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112438 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register